## The Effect of Different Intra-articular Injections on Pain and Function in Primary Gonarthrosis

01.04.2020

Dear Volunteer,

This research, "The effect of different intra-knee injection preparations on pain and functional activity in primary gonarthrosis", was conducted by Dr.Mahmut Enes Kayaalp. The study was planned to compare the types of treatment modalities in patients with knee osteoarthritis. The pain in knee is generated from the 'calcification' which leads the malfunctioning of the joint. With the results to be obtained from your answers, the effectiveness of the treatments applied and thus the treatments to be applied from now on can be planned. Therefore, it is very important that you answer all of the questions. Some drug reactions may develop in oral and local treatment. These can be counted as an mild allergic reaction such as gastritis or rash. In addition, low rates of complications can be seen in intra-knee injections. These are, development of infection in the knee joint, the development of an allergic reaction, and the formation of a rash on the skin. In such a case, the contact information is shared below so that you can reach the doctor who administers the treatment.

Your participation in the research is on a voluntary basis. Information obtained through this form will remain confidential and will only be used for research purposes (or "scientific purposes"). You can choose not to participate in the study, or if you do not want to fill out the questionnaire, you can terminate it.

Do not write your name and surname on the questionnaire.

Our survey consists of 2 parts. Eleven questions, 5 minutes. In this study, which will take your time, indicate your answers by ticking the appropriate option among the options next to the questions. Also, mark your visual pain score shown to you by choosing the score you think is appropriate. You can only give one answer to each of the questions. Thank you for answering the survey.

If you have any questions about the study, you can contact the following person(s):

Dr.Mahmut Enes Kayaalp 0536 515 7274

Dr. Yiğit Umur Cırdı 0535 3540999